CLINICAL TRIAL: NCT06684067
Title: A Prospective Randomized Controlled Trial to Evaluate the Effect of Patient Navigation on Colonoscopy Screening Rate for Colorectal Cancer (CRC) in University Malaya Medical Centre (UMMC)
Brief Title: Effect of Patient Navigation on Colonoscopy Completion Screening Rate for Colorectal Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: MREC ID No: 202057-8603
Record Dates: First submitted 2024-10-04; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer Screening; Patient Navigation
Keywords: RCT; colorectal cancer screening; patient navigation; Malaysia; depression; anxiety; HADS; GHQ12
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient navigation (Experimental): Participants in the intervention arm will undergo a patient navigation process
  Interventions: Behavioral: Patient navigation
- No navigation (No Intervention): Participants in the control arm will receive standard instructions and not undergo the patient navigation process.

INTERVENTIONS:
Behavioral: Patient navigation — Participants will receive online educational material, hospital site navigation guidance and direct contact with the patient navigator, in addition to standard instructions on the colonoscopy procedure.
  Arms: Patient navigation

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of patient navigation on colonoscopy completion rates in a population screened for colorectal cancer. The main question[s] it aims to answer are:

Are colonoscopy completion rates in colorectal cancer screening increased in navigated (intervention arm) compared with non-navigated (control arm) participants?

Is mental well-being, as measured by HADs and GHQ12 scores, better in the intervention arm compared with the control arm?

Participants in the intervention arm will receive:

* standard clinic instructions for the colonoscopy
* phone calls from the patient navigator to discuss the purpose, preparation, and additional information regarding the colonoscopy procedure
* a webpage QR code consist of information on visual image on colonoscopy preparation and procedures, layout and map guidance to navigate in the hospital
* a direct line for phone calls to patient navigators for further guidance on overcoming barriers

Participants in the control arm will only receive:

* standard clinic instructions for the colonoscopy
* one phone call from the patient navigator to discuss the colonoscopy procedure

ELIGIBILITY:
Inclusion Criteria:

* Average risk for CRC
* More than 50 years of age
* Capacity for informed consent
* IFOBT positive

Exclusion Criteria:

* Moderate or high risk CRC
* Previous CRC screening
* Symptomatic

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Colonoscopy completion rate | 90 days
  The numerator in both arms comprises participants who successfully attended and underwent colonoscopy within 90 days of recruitment. The denominator in both arms comprises all participants randomized to that arm. Colonoscopy completion rate was defined as the percentage of participants who completed colonoscopy within 90 days of randomization.

SECONDARY OUTCOMES:
Mental health - anxiety and depression | 90 days
  The mental health of participants in both arms was assessed pre- and post-colonoscopy using the Hospital Anxiety & Depression Scale (HADS). The score may range from 0-21. Scores of 0-7 are normal, 8-10 is mild, 11-14 is moderate and 15-21 is severe anxiety or depression.
Mental health - General psychological distress | 90 days
  The mental health of participants in both arms was assessed pre- and post-colonoscopy using the General Health Questionnaire 12 (GHQ12) tool as a measure of general psychological distress. Each item in the 12-item questionnaire was scored on a Likert scale of 0-3, for a total score ranging from 0-36. High scores indicate worse health.

CONTACTS AND LOCATIONS:
Overall Officials: April C Roslani, Master of Surgery, Principal Investigator — Universiti Malaya
Locations (1):
- Faculty of Medicine, Universiti Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Informed consent was only given for the purposes of this study.